CLINICAL TRIAL: NCT06932380
Title: A Talus Implant in Patients Between 20-60 Years of Age Followed up for a Minimum of 2 Years After Surgery: A Pilot Study
Brief Title: A Talus Implant in Patients Between 20-60 Years of Age Followed up for a Minimum of 2 Years After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/09300-3
Record Dates: First submitted 2025-03-31; First posted 2025-04-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cartilage Lesion
Keywords: focal cartilage injury; ankle cartilage; patient-specific implant; pilot study

STUDY DESIGN:
Intervention Model Description: This interventional pilot study employs a prospective cohort design to evaluate the safety, feasibility, and efficacy of the patient-specific Episurf Episealer talus implant in treating osteochondral lesions of the ankle. Ten patients aged 20 to 60 years with symptomatic cartilage defects unresponsive to conservative or prior surgical treatment will be included. The intervention consists of open surgical implantation of a custom-made cobalt-chromium implant tailored to each patient's joint anatomy. Outcomes will be assessed through clinical function scores (AOFAS), pain and satisfaction measures (NRS), and health-related quality of life (EQ-5D-5L) over a two-year follow-up period. The study aims to provide preliminary evidence on the implant's clinical performance, with revision rates and complications as primary endpoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talus prosthesis (Experimental): This study consists of a single-arm intervention evaluating the Episurf Episealer talus implant in patients with symptomatic osteochondral lesions of the ankle. All included patients will undergo open surgical implantation of the patient-specific cobalt-chromium implant, designed to restore joint congruency and improve function. Standardized postoperative care, including rehabilitation and follow-up assessments at 6 weeks, 6 months, 1 year, and 2 years, will be provided. Primary outcomes include revision rate and complication incidence, while secondary measures assess pain, functional improvement, and health-related quality of life.
  Interventions: Procedure: Talus prosthesis

INTERVENTIONS:
Procedure: Talus prosthesis — The Episealer Talus is an individualised resurfacing implant intended for use on either the medial or lateral talus. It aims to treat patients suffering from pain and reduced mobility due to focal osteochondral lesions in the talus.

SUMMARY:
The project will investigate safety, feasibility and efficiency when using Episurf Episeal talus implant in patients with osteochondral ankle injuries. Assessments includes revision rate, complications, pain, function and quality of life over two years. Ten patients (aged 20-60) who have not responded to previous treatment will participate based on informed and written consent. The project uses a prospective cohort design where the patients receive a customized surgical procedure. Data on clinical function, pain and patient satisfaction collected using the AOFAS ankle score, NRS and EQ-5D-5L questionnaire at 6 weeks, 6 months, 1 year and 2 years after the operation. The study can provide valuable insight into the treatment of ankle osteoarthritis, improve the patient's quality of life and function, and represent a step forward in orthopedic surgery, especially for younger, active patients. The results are shared with it the medical community and the general public through publications and presentations.

DETAILED DESCRIPTION:
Localized cartilage injuries in the ankle occur when distinct areas of the cartilage in the ankle joint become damaged or worn down. This can lead to pain, swelling, reduced mobility and function, and an increased risk of osteoarthritis over time. The challenge with these injuries is that cartilage has a limited capacity for self-healing due to its lack of direct blood supply. Treatment options remain limited, as conventional methods such as physiotherapy or anti-inflammatory medications only address symptoms rather than the underlying damage. More invasive procedures, such as joint replacement or extensive reconstructive surgery, are associated with prolonged rehabilitation periods and variable success rates, particularly in younger, active patients. This highlights the need for precise, customized treatment solutions that can directly repair the damage and effectively restore joint function. A patient-specific implant has been designed to address focal cartilage injuries in joints, primarily in the knee but also in the ankle. The implant is based on advanced imaging and 3D modeling to adapt to the patient's unique joint anatomy and extent of injury. The method involves open surgery to replace the damaged cartilage and adjacent bone with a metal implant (cobalt-chromium) that mimics the patient's original joint surface. This facilitates targeted pain relief and improved joint function, offering a personalized treatment alternative for patients with localized cartilage defects. Compared to traditional ankle joint replacements or arthrodesis, the use of this implant is considered less invasive and associated with a shorter recovery period, reducing patient burden and allowing for a quicker return to daily activities. Additionally, the patient-specific design of the implant has the potential to minimize implant-related complications, such as implant wear and implant-related pain. Early clinical studies on this implant have shown promising results regarding pain relief, improved joint function, and patient satisfaction. However, only a limited number of reports exist to date, and further studies are needed to assess the long-term effects of the implant on pain, function, and quality of life.

The implant may represent a significant advancement in orthopedic surgery and has the potential to improve the quality of life for patients suffering from ankle joint injuries and osteochondral lesions.

In conjunction with the introduction of this method and implant, particularly in younger patients, the investigators aim to conduct a pilot study on the early outcomes of the first ten patients, focusing on safety, feasibility, and efficacy.

This project aims to evaluate the surgical outcomes in patients aged 20 to 60 years with challenging cartilage injuries in the ankle, two years postoperatively following implantation of a custom-made talus implant. The study focuses on safety, feasibility, and efficacy. Complications and adverse events will be recorded.

Clinical function will be assessed using the American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score, a well-validated and reliable scoring system, while HRQoL will be assessed using the EQ-5D-5L score.

Ten patients with osteochondral lesions will be included in the study. Patients will be selected from a clinical population with moderate to severe symptoms and will be treated at an orthopedic clinic (DS) with expertise in managing ankle osteoarthritis/cartilage injuries and performing the talus implant implantation. Through this recruitment process, the investigators aim to establish a cohort that reasonably reflects the patient population with ankle osteoarthritis at our clinic, thereby enhancing the quality and relevance of the research.

Upon inclusion, patients will undergo a clinical examination, X-ray, and MRI imaging of the foot to assess the extent of the injury and joint geometry. The Berndt-Harty classification system will be used to categorize the injury based on radiographic images, and the Bristol-Hepple classification will be employed to describe lesion size, edema, displacement, and cyst formation based on MRI images. Patients will undergo implantation of the talus implant performed by a qualified orthopedic surgical team. Pre- and postoperative pain management protocols will be implemented. Standard postoperative follow-up plans, including rehabilitation and physiotherapy, will be provided. Patients will be followed up clinically at 6 weeks, 6 months, 1 year, and 2 years postoperatively.

Additional data collected include: Demographic data: Age, sex, surgical time (minutes).

Clinical data: Time of diagnosis, treatment initiation, treatment type, and treatment course.

Patients will be informed about the study and will provide written consent before inclusion. To ensure ethical and legal informed consent, patients will receive a detailed consent form explaining the nature of the study, what participation entails, and how patient data will be managed to protect confidentiality. Only after obtaining written consent will patients be included in the study.

In this study, the power calculation is challenged by a limited patient sample, which affects the potential for statistical significance. With a single cohort of 10 patients over a two-year period, the sample size restricts the ability to detect statistically significant differences in AOFAS and EQ-5D-5L scores. Reduced statistical power is an inherent consequence of the small sample size. The results, primarily descriptive and exploratory, must be interpreted with caution and regarded as a foundation for further research. Alternative analytical approaches will be considered to maximize the value of the collected data.

The following data processing and statistical analysis methods are planned:

* Descriptive statistics to summarize demographic and baseline clinical characteristics of participants.
* T-tests or Wilcoxon signed-rank tests to compare pre- and postoperative outcomes on continuous variables such as pain (NRS), AOFAS scores, and HRQoL (EQ-5D-5L), depending on data distribution.
* ANOVA or Kruskal-Wallis tests for comparisons across multiple time points or groups.
* Linear regression models to analyze relationships between predictors (e.g., age, sex, injury severity) and outcome variables (e.g., pain, function, HRQoL).
* Calculation of the Minimum Clinically Important Difference (MCID) for EQ-5D-5L to establish the smallest score change perceived as clinically meaningful by patients.
* Kaplan-Meier survival analysis to estimate revision rates over time.
* Cox proportional hazards models to assess risk factors for potential implant revisions. A detailed analysis plan will be developed before data collection begins to ensure that the study has sufficient power to detect any significant differences or associations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-60 years with symptomatic osteochondral lesions of the ankle where conservative treatment or previous surgery has been unsatisfactory.
* Patients with a limited cartilage defect that qualifies for Episealer implantation.
* Patients who have provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients with an active infection in the ankle.
* Patients with extensive cartilage damage where Episealer is not indicated.
* Patients with osteoarthritic changes on the tibial side of the ankle joint.
* Patients with severe joint instability.
* Patients with severe neurological or systemic diseases.
* Patients who smoke.
* Patients with substance abuse issues.
* Patients unable to attend follow-ups due to distance or other factors.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients undergoing revision surgery | From the time of the index surgery throughout the entire 24-month follow-up period.
  Revision surgery involves replacing or removing part or all of the talus prosthesis. This may be necessary in the event of various problems with the prosthesis, for example that the prosthesis has loosened from the bone, wear of the prosthesis materials, infection or if the prosthesis dislocates.

SECONDARY OUTCOMES:
Patient satisfaction on a scale from 0 to 10 | Baseline - from the time of the index surgery - throughout the entire 24-month follow-up period.
  Patient satisfaction is assessed by the use of NRS, or Numerical Rating Scale, which is a widely used method for assessing patients' experience of satisfaction. It consists of a scale from 0 to 10, where 0 represents or "completely dissatisfied" and 10 indicates "completely satisfied".
  Patients are asked to rate their satisfaction level by selecting a number that best describes their current condition.
  The NRS is easy to administer and understand, and can be used in a number of medical and research contexts to quantify degree of satisfaction.
  This method is particularly useful for following changes in the patient's condition over time, as well as evaluating the effect of treatments or interventions. In assessments of satisfaction, the person answers a standard question from the project staff. The NRS has been found to be both reliable and valid and is widely used when assessing satisfaction.
Patient pain on a scale from 0 to 10 | Baseline - from the time of the index surgery - throughout the entire 24-month follow-up period.
  Pain is assessed by the use of NRS, or Numerical Rating Scale, which is a widely used method for assessing patients' experience of pain. It consists of a scale from 0 to 10, where 0 represents "no pain" and 10 indicates "worst imaginable pain".
  Patients are asked to rate their pain level by selecting a number that best describes their current condition.
  The NRS is easy to administer and understand, and can be used in a number of medical and research contexts to quantify pain intensity. This method is particularly useful for following changes in the patient's condition over time, as well as evaluating the effect of treatments or interventions. In assessments of pain, the person answers a standard question from the project staff. The NRS has been found to be both reliable and valid and is widely used when assessing pain.
AOFAS ankle score on a scale from 0 to 100 | Baseline - from the time of the index surgery throughout the entire 24-month follow-up period.
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Rating System is a standardized evaluation of the clinical status of the ankle-hindfoot. It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion. Scores range from 0 to 100, with healthy ankles receiving 100 points.
  This score may be used to assess the ankle, subtalar, talonavicular, and calcaneocuboid joint levels and may be useful for fractures, arthroplasty, arthrodesis, and instability procedures.
EQ-5D-5L score | Baseline - from the time of the index surgery - throughout the entire 24-month follow-up period.
  The EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version) is a generic tool for Patient-Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease.
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Drammen Sykehus, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is not prohibited by the Ethics Committee and will thus not be done.